CLINICAL TRIAL: NCT04460677
Title: ASD (Autism Spectrum Disorder) Telehealth for Distress Related to COVID-19 (Coronavirus Disease)
Brief Title: ASD (Autism Spectrum Disorder) Telehealth for Distress Related to COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Vanessa H. Bal, PhD, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro2020001593
Record Dates: First submitted 2020-07-06; First posted 2020-07-07 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Psychological Distress; Stress, Psychological; Autism Spectrum Disorder
Keywords: smartphone; ecological momentary intervention (EMI); ecological momentary assessment (EMA)
MeSH Terms: conditions — Stress, Psychological; Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional Support Plan (ESP) + Weekly Monitoring (Experimental): This will involve weekly assessments without prompting to use the plan.
  Interventions: Behavioral: Emotional Support Plan
- Emotional Support Plan (ESP) + 4x Daily Monitoring (Experimental): Participants in this arm will be prompted on their phones 4x/day randomly, to report on activities, mood, suicidal ideation, distress level and ESP use since the last prompt
  Interventions: Behavioral: Emotional Support Plan; Behavioral: Daily Monitoring

INTERVENTIONS:
Behavioral: Emotional Support Plan — The Emotional Support Plan (ESP) is designed to help adults to cope during periods of acute distress, such as those experienced during the COVID-19 pandemic.
Behavioral: Daily Monitoring — The daily monitoring will remind participants 4x/day to report on their mood, distress, etc. and use their ESP if needed.
  Arms: Emotional Support Plan (ESP) + 4x Daily Monitoring

SUMMARY:
The purpose of this study is to evaluate the feasibility, acceptability and effectiveness of a brief, telehealth intervention (the Emotional Support Plan), intended to support autistic adults to cope with their negative emotions during and/or after the COVID-19 pandemic. The first objective is to develop and refine a brief telehealth-delivered treatment, the Emotional Support Plan (ESP), to help promote adults to cope during periods of acute distress, such as those experienced during the COVID-19 pandemic. The second objective is to assess the feasibility and effectiveness of the ESP to support autistic adults to implement emotion regulation strategies during periods of acute distress. The last objective is to yield preliminary data to apply for extramural grants to validate these methods to monitor and support mental health of autistic adults during key transitions (e.g., starting college).

ELIGIBILITY:
Inclusion Criteria Adults 18 years or older with previously established diagnoses in ASD will be invited to participate. Adults who have a verbal IQ above 70 or who are students admitted to a college or university will be included in the study.

Exclusion Criteria

* Individuals who are younger than 18 years old or who does not have diagnosis of ASD will excluded from the study as the purpose of the current research is to evaluate the validity of ESPs in adults with autism.
* Adults who are unable to understand English will be excluded because the instruments being investigated are currently only validated in English and the study team is not sufficiently fluent in other languages to provide assurance that informed consent could be obtained (or intervention provided) in a language besides English.
* Subjects without access to a compatible iOS and Android smartphone (nearly all phones from the past 10 years are compatible) will be excluded because the study requires subjects to record responses on a smartphone app. Individuals will not be excluded from the study based on race, ethnicity or gender.
* Subjects who have a verbal IQ below 70 will be excluded as this is a study that requires self-report and engagement in a one-on-one intervention.
* If the PI's clinical judgment is that it would not be in the adult's best interest to be enrolled, they may also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
Decreased distress on Patient Health Questionnaire (PHQ-9) | 8 week study period
  The PHQ-9, assessed weekly, is a 9-item questionnaire of psychological function over the past week with all items on a "0" (not at all) to "3" (nearly every day) scale. Higher scores equal more distress.
Decreased distress on EMA reports | 8 week study period
  EMA (Ecological Momentary Assessment) reports of decreased distress (in ESP + daily monitoring group only). Higher scores on the item equal higher levels of distress.
Decreased anxiety symptoms on the Generalized Anxiety Disorder Questionnaire (GAD-7) | 8 week study period
  The GAD-7, assessed weekly, is a 7-item questionnaire of anxiety symptoms over the past week with all items on a "0" (not at all) to "3" (nearly every day) scale. Higher scores equal more anxiety.

SECONDARY OUTCOMES:
Adult Self Report (ASR) | 8 week study period
  The ASR is a measure of adaptive functioning and psychopathology (e.g., anxiety, depression symptoms). Most of the items are on a 3 point scale including: (0) Not true, (1) Somewhat or sometimes true, and (2) Very often or often true.

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers University, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No